CLINICAL TRIAL: NCT06984809
Title: Evaluation of the Invest in Play Program - a New Parent Intervention for Children With Problem Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: NORCE Norwegian Research Centre AS (Other); NTNU Health (sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/785387; 2025-957314 (Other: Norwegian Agency for Shared Services in Education and Research (SIKT))
Record Dates: First submitted 2025-05-09; First posted 2025-05-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-09

CONDITIONS: Problem Behavior; Attention Deficit and Disruptive Behavior Disorders
Keywords: parent intervention; parent practices; emotion regulation; parent-child relationship; parental attributions
MeSH Terms: conditions — Problem Behavior; Attention Deficit and Disruptive Behavior Disorders; Emotional Regulation | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control condition will receive usual care, e.g., further assessments, school meetings, individual care and/or psycho education.
- Invest in Play group (Experimental): Intervention group receiving Invest in Play (iiP), a 12 session program provided weekly to parents with children with problem behavior.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — The intervention group will receive Invest in Play (iiP), a 12 session group-based parent program, which is led by two trained group leaders.
  Other Names: Invest in Play (iiP)
  Arms: Invest in Play group

SUMMARY:
The goal of this clinical trial is to test if the invest in Play (iiP) parent program can reduce problem behaviors in children and improve parenting practices in families with children who show challenging behaviors. The main questions it aims to answer is:

• Does the iiP program reduce children's problem behaviors?

Researchers will compare families in the iiP program to families in a control group to see if the program leads to better outcomes for children and parents.

Participants will be randomly assigned to either the iiP program group or the control group and complete surveys before and after the program to see if iiP is reducing children's problem behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children between 6-12 years of age referred to out-patient clinics for treatment of behavioural problems.
* Children scoring above a pre-defined mean cut off score (over the 90 percentile) on the Eyberg Child Behavior Inventory (ECBI; Eyberg & Ross, 1978) based on Norwegian norms (Reedtz et al., 2008), as reported by parents.

Exclusion Criteria:

- Severe developmental delay (in children or parents), autism spectrum disorder, inability to understand Norwegian, or other reasons why the parent(s) are not expected to benefit from group therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Eyberg Child Behavior Inventory (ECBI) score at different time points (from baseline up to 12 weeks). | From baseline to the end of treatment at 12 weeks.
  Child problem behavior will be measured using the Eyberg Child Behavior Inventory (ECBI), where the change score from baseline to 12 weeks post intervention is the primary outcome. The measure consists of 36 items, which is scored on parents' notion about the intensity (1 = never to 7 = always), and whether child behavior is a problem (0 = no and 1 = yes, range 0-36). A total score is calculated, ranging from range 36-252. High intensity scores indicate more intense problems, and a high problem score indicate a higher frequency of problem behaviors. The ECBI has demonstrated strong internal consistency, test-retest reliability, and discriminant validity and has been shown to be a sensitive indicator of intervention efficacy for child behavior problems.

SECONDARY OUTCOMES:
Change in the Social Competence Scale-Parent (SCS-P) score at different time points (from baseline up to 12 weeks). | From baseline to the end of treatment at 12 weeks.
  Social Competence Scale-Parent (SCS-P) is a 12-item measure for assessing two domains of children's social competence, namely prosocial skills ("Your child can give suggestions and opinions without being bossy") and emotion regulation (e.g., "Your child can calm down when excited or all wound up."). The items are rated on a scale from 0 = "Not at all" to 4 = "Very well". For this study, the emotion regulation skills subscale (6 items) will be used, and the subscale is scored as a mean of responses, where higher scores indicate better emotion regulation.
Change in the Kidscreen-10 score at different time points (from baseline up to 12 weeks). | From baseline to the end of treatment at 12 weeks.
  Kidscreen-10 index parent version measures children's health related global quality of life (HRQoL). The 10-item version is the short version of the KIDSCREEN-52 and KIDSCREEN-27 instrument and is rated on a scale from 1 = "Not at all" to 5 = "to a large extent". A total score is calculated, where higher scores indicates better HRQoL.
Change in Strengths and Difficulties Questionnaire (SDQ) score at different time points (from baseline up to 12 weeks). | From baseline to the end of treatment at 12 weeks.
  The Strength and Difficulties Questionnaire (SDQ) is a brief behavioral screening questionnaire consisting of 25 items, divided by on 5 subscales (prosocial, hyperactivity, emotional symptoms, conduct problems and peer problems), scored from 0 = not true, 1 = somewhat true and 2 = certainly true. The parent version will be used in this study. A total score from each subscale is calculated. In addition, the last four subscales are added together to generate a total difficulties score (based on 20 items), where a higher score indicate more difficulties.
Change in the Parenting and Family Adjustment Scales (PAFAS) score at different time points (from baseline up to 12 weeks). | From baseline to the end of treatment at 12 weeks.
  Parenting and Family Adjustment Scales (PAFAS) is a 40-item measure assessing parent and family functioning through five domains (parenting practices, quality of parent-child relationship, parental emotional adjustment, positive family relationships, and parental teamwork), which are all considered to be important for child outcomes. The items are rated on a 4-point scale from 0 = not true for me at all to 3 = true of me very much. The scores are summed (some scores are reversed), where higher scores indicate a more dysfunctional family life.
Change in the Parent Stress Scale (PSS) scores at different time points (from baseline up to 12 weeks). | From baseline to the end of treatment at 12 weeks.
  The Parent Stress Scale (PSS) is an 18-item questionnaire assessing parents' feelings about their parenting role, exploring both positive aspects (e.g. emotional benefits, personal development) and negative aspects of parenthood (e.g. demands on resources, feelings of stress). The scale is rated on a 5-point scale from 1 = Strongly disagree to 5 = Strongly agree. Some of the scores are reversed, and a total score is calculated. A high score indicate high stress levels. We will use the subscale with six items addressing parent stress and the more negative aspects of parenthood in this study.
Change in the Parent Cognition Scale (PCS) score at different time points (from baseline up to 12 weeks). | From baseline to the end of treatment at 12 weeks.
  The Parent Cognition Scale (PCS) is a 16-item self-report measure of parental attributions of child behavior. The scale consists of two subscales, which assesses child-responsible attributions (e.g., "I'm not structured enough with my child") and parent-causal attribution (e.g., "I'm not structured enough with my child"). The items are rated on a scale from 0 = always true to 5 = never true, all being reverse scored. This means that higher scores indicate more negative attributions.
Change in the Me as parent - Short form (MaaPs-SF) score at different time points (from baseline up to 12 weeks). | From baseline to the end of treatment at 12 weeks.
  Me as parent - Short form (MaaPs-SF) is a four-item measure to assess parent self-efficacy. The scale is derived from the original 16-item version (Hamilton et al., 2014), developed to assess parenting self-regulation. The MaaPs-SF is rated on a 5-point scale from 1 = Strongly disagree to 5 = Strongly agree. The four items are added to provide a total score, where a higher score indicates better parenting self-efficacy.
Change in the Parental Emotion Regulation Inventory (PERI-2) score at different time points (from baseline up to 12 weeks). | From baseline to the end of treatment at 12 weeks.
  The Parental Emotion Regulation Inventory (PERI-2) is a 23-item self-report measure to assess parents own self-regulation. The items consist of different emotion regulation strategies which are rated on a 7-point scale ranging from 1 (I never do this) to 7 (I very often do this), comprising four different subscales (Reappraisal, Suppression, Escape and Capitulation). A score for each subscale is calculated, where a high score indicate that the strategies within that factor are more used.

OTHER OUTCOMES:
Change in Eyberg Child Behavioral Inventory (ECBI) score from post-intervention to three months follow up. | From post-treatment to three months post intervention.
  Investigators want to assess whether the scores changes in the Invest in Play intervention group three months post intervention.
  The Eyberg Child Behavioral Inventory (ECBI) is a well-validated measure for evaluating child problem behavior. The measure consists of 36 items, which is scored on parents' notion about the intensity (1 = never to 7 = always), and whether child behavior is a problem (0 = no and 1 = yes, range 0-36). A total score is calculated, ranging from range 36-252. High intensity scores indicate more intense problems, and a high problem score indicate a higher frequency of problem behaviors.
Change in the Social Competence Scale-Parent (SCS-P) score from post-intervention to three months follow up. | From post-treatment to three months post intervention.
  Investigators want to assess whether the scores changes in the Invest in Play intervention group three months post intervention.
  The Social Competence Scale-Parent (SCS-P) is a 12-item measure for assessing two domains of children's social competence, namely prosocial skills ("Your child can give suggestions and opinions without being bossy") and emotion regulation (e.g., "Your child can calm down when excited or all wound up."). The items are rated on a scale from 0 = "Not at all" to 4 = "Very well". For this study, the emotion regulation skills subscale (6 items) will be used, and the subscale is scored as a mean of responses, where higher scores indicate better emotion regulation.
Change in Kidscreen-10 score from post-intervention to three months follow up. | From post-treatment to three months post intervention.
  Investigators want to assess whether the scores changes in the Invest in Play intervention group three months post intervention.
  Kidscreen-10 index parent version measures children's health related global quality of life (HRQoL). The 10-item version is the short version of the KIDSCREEN-52 and KIDSCREEN-27 instrument and is rated on a scale from 1 = "Not at all" to 5 = "to a large extent". A total score is calculated, where higher scores indicates better HRQoL.
Change in Strengths and Difficulties Questionnaire (SDQ) score from post-intervention to three months follow up. | From post-treatment to three months post intervention.
  Investigators want to assess whether the scores changes in the Invest in Play intervention group three months post intervention.
  The Strength and Difficulties Questionnaire (SDQ) is a brief behavioral screening questionnaire consisting of 25 items, divided by on 5 subscales (prosocial, hyperactivity, emotional symptoms, conduct problems and peer problems), scored from 0 = not true, 1 = somewhat true and 2 = certainly true. The parent version will be used in this study. A total score from each subscale is calculated. In addition, the last four subscales are added together to generate a total difficulties score (based on 20 items), where a higher score indicate more difficulties.
Change in the Parenting and Family Adjustment Scales (PAFAS) from post-intervention to three months follow up. | From post-treatment to three months post intervention.
  Investigators want to assess whether the scores changes in the Invest in Play intervention group three months post intervention.
  Parenting and Family Adjustment Scales (PAFAS) is a 40-item measure assessing parent and family functioning through five domains (parenting practices, quality of parent-child relationship, parental emotional adjustment, positive family relationships, and parental teamwork), which are all considered to be important for child outcomes. The items are rated on a 4-point scale from 0 = not true for me at all to 3 = true of me very much. The scores are summed (some scores are reversed), where higher scores indicate a more dysfunctional family life
Change in the Parent Stress Scale (PSS) from post-intervention to three months follow up. | From post-treatment to three months post intervention.
  Investigators want to assess whether the scores changes in the Invest in Play intervention group three months post intervention.
  The Parent Stress Scale (PSS) is an 18-item questionnaire assessing parents' feelings about their parenting role, exploring both positive aspects (e.g. emotional benefits, personal development) and negative aspects of parenthood (e.g. demands on resources, feelings of stress). The scale is rated on a 5-point scale from 1 = Strongly disagree to 5 = Strongly agree. Some of the scores are reversed, and a total score is calculated. A high score indicate high stress levels. We will use the subscale with six items addressing parent stress and the more negative aspects of parenthood in this study.
Change in the Parent Cognition Scale (PCS) score from post-intervention to three months follow up. | From post-treatment to three months post intervention.
  Investigators want to assess whether the scores changes in the Invest in Play intervention group three months post intervention.
  The Parent Cognition Scale (PCS) is a 16-item self-report measure of parental attributions of child behavior. The scale consists of two subscales, which assesses child-responsible attributions (e.g., "I'm not structured enough with my child") and parent-causal attribution (e.g., "I'm not structured enough with my child"). The items are rated on a scale from 0 = always true to 5 = never true, all being reverse scored. This means that higher scores indicate more negative attributions.
Change in the Me as parent - Short form (MaaPs-SF) score from post intervention to three months follow up. | From post-treatment to three months post intervention.
  Investigators want to assess whether the scores changes in the Invest in Play intervention group three months post intervention.
  Me as parent - Short form (MaaPs-SF; Matthews, et al., 2022) is a four-item measure to assess parent self-efficacy. The scale is derived from the original 16-item version (Hamilton et al., 2014), developed to assess parenting self-regulation. The MaaPs-SF is rated on a 5-point scale from 1 = Strongly disagree to 5 = Strongly agree. The four items are added to provide a total score, where a higher score indicates better parenting self-efficacy.
Change in the Parental Emotion Regulation Inventory (PERI-2) from post intervention to three months follow up. | From post-treatment to three months post intervention.
  Investigators want to assess whether the scores changes in the Invest in Play intervention group three months post intervention.
  The Parental Emotion Regulation Inventory (PERI-2) is a 23-item self-report measure to assess parents own self-regulation. The items consist of different emotion regulation strategies which are rated on a 7-point scale ranging from 1 (I never do this) to 7 (I very often do this), comprising four subscales (Reappraisal, Suppression, Escape and Capitulation). A score for each subscale is calculated, where a high score indicate that the strategies within that factor are more used.

CONTACTS AND LOCATIONS:
Overall Officials: Lene-Mari P. Rasmussen, Ph.d, Principal Investigator — UiT The Arctic University of Norway
Locations (4):
- Norway (4):
  - Haukeland university hospital, department of mental health care for children and adolescents, Bergen
  - Helse Fonna HF, BUP Stord, Haugesund
  - Helse Nord-Trøndelag HF, Barne- og ungdomspsykiatrisk avdeling (BUP), Namsos
  - OUS/PHA/BUPA/BUP Oslo Nord, Oslo

IPD SHARING:
Plan to Share IPD: Yes
De-identified data (data where personal identifying characteristics have been removed) may be shared with national or international collaborators in Denmark and the Netherlands for use in comparative studies. This primarily applies to information related to the child's behavior, parental stress, and user satisfaction.
  Data from the study can also be made available for other researchers upon request (see details below under access criteria).
Supporting Information: ICF
Time Frame: 31.12.2028-31.12.2033.
Access Criteria: Reasearcher affiliated to recognized academic institutions can request access by taking contact with a proposal that describes planned analyses must be submitted and will be evaluated by the project leader and data manager.